CLINICAL TRIAL: NCT05453149
Title: Piloting an Online Integrated Behaviour Change and Physical Activity Program for Those With Neurological Conditions
Brief Title: Piloting an Online Integrated Behaviour Change and Physical Activity Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 121214
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Neurological Disorder; Behavioural Change Intervention; Physical Activity
MeSH Terms: conditions — Nervous System Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persons with Neurological Conditions (Experimental)
  Interventions: Behavioral: Integrated Physical Activity and Behavioural Change Intervention

INTERVENTIONS:
Behavioral: Integrated Physical Activity and Behavioural Change Intervention — Physical Activity (PA) Component: A group-based PA program geared to the level of injury and mobility delivered through web conferencing software. Participants select at three sessions weekly over 10 weeks. Sessions include 45 mins of exercise (i.e boxercise; aerobics; yoga) and 15 mins of social interaction with the group.
  Behavioural Change Component: Participants will also receive synchronous 1:1 sessions (approximately 20 mins/week) with a trained clinician on behavioural strategies to initiate and maintain engagement in PA over the 10-week period. Content of the sessions includes: providing information on PA and the self-management of impairments and related symptoms; evaluating barriers to engagement (e.g. fear of injury); and behavioural strategies.

SUMMARY:
There is a significant disparity in access to physical activity programs for people with mobility impairments, which greatly impacts mobility, function and long-term wellbeing. This study will test an online, group-based intervention consisting of exercise and behaviour activation strategies targeting these and other outcomes. Importantly, this programming will be applied to patient groups across several clinical programs at Parkwood Institute.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over
* Neurological condition (i.e., brain injury, stroke)
* Completed rehabilitation and living in the community
* Participants must have some upper limb function permitting arm movement against gravity
* Physician clearance to participate in the study.

Exclusion Criteria:

* Not cleared by a physician.
* Not able to move upper limbs against gravity.
* No internet access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Self Efficacy | baseline, 10 weeks, 3 months
  Self-Efficacy for Managing Chronic Disease 6-item Scale; Scale for the assessement of phase-specific self-efficacy of physical activity
Change in Physical Activity | baseline, 10 weeks, 3 months
  Physical Activity scale for individuals with physical disabilities (PASIPD)
Change in Life Participation | baseline, 10 weeks, 3 months
  NeuroQoL ability to participate; NeuroQoL satisfaction with participation
Change in health behaviour | baseline, 10 weeks, 3 months
  Scale for assessment of implementation planning and coping planning
Change in fear of falls | baseline, 10 weeks, 3 months
  Falls Efficacy Scale - International
Change in exercise expectations | baseline, 10 weeks, 3 months
  Outcome Expectations for Exercise scale
Change in Mood | baseline, 10 weeks, 3 months
  PHQ9
Change in Anxiety | baseline, 10 weeks, 3 months
  GAD7
Change in personality | baseline, 10 weeks, 3 months
  BFI/AAQ

CONTACTS AND LOCATIONS:
Overall Officials: Swati Mehta, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's